CLINICAL TRIAL: NCT01086969
Title: Safety and Immunogenicity Study for Use of Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra®) in Healthy Subjects 2-55 Years of Age in India
Brief Title: A Study of Meningococcal Vaccine, Menactra® in Healthy Subjects in India
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA51; UTN: U1111-1111-5608 (Other: WHO)
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Results first posted 2012-02-03 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Meningococcal Infection; Meningitis
Keywords: Meningococcal Infection; Meningitis, Bacterial; Menactra®
MeSH Terms: conditions — Meningococcal Infections; Meningitis; Meningitis, Bacterial | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): Participants in three age cohorts - Children: 2 - 11 years of age; Adolescents: 12 - 17 years of age, and Adults: 18 - 55 years of age will be enrolled.
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate (Menactra®)

INTERVENTIONS:
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate (Menactra®) — 0.5 mL, Intramuscular
  Other Names: Menactra®

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of a single dose of Menactra® vaccine to support registration.

Primary Objectives:

* To describe the antibody titers measured by serum bactericidal activity using baby rabbit complement (SBA-BR) before and after Menactra® vaccination.
* To describe the safety profile of participants after one dose of Menactra®.

DETAILED DESCRIPTION:
Participants will be enrolled in three age cohorts: Children: 2 - 11 years of age; Adolescents: 12 - 17 years of age, and Adults: 18 - 55 years of age to receive a single dose of Menactra®. They will be followed for a duration of 30 days after vaccination.

ELIGIBILITY:
Inclusion Criteria :

* Aged 2 to 11 years or Aged 12 to 17 years or Aged 18 to 55 years of age on the day of inclusion
* For participants aged 2 to 11 years: Provision of informed consent form signed by the parent(s) or legal representative.
* For participants aged 12 to 17 years: Provision of assent form signed by the participant and informed consent form signed by the parent(s) or legal representative.
* For participants aged 18 to 55 years: Provision of informed consent form signed by the participant. If the participant or the participant's parents or legally accepted representative (participants aged 2 to 17 years) are illiterate, an independent witness is required to sign the consent form.
* Participant and parent/legally acceptable representative (if applicable) able to attend all scheduled visits and comply with all trial procedures
* For a woman of child-bearing potential, sexually active, use of a medically acceptable and effective method of contraception for at least 4 weeks prior to vaccination, until at least 4 weeks after vaccination (not applicable for participants aged 2 to 17 years' females not of child-bearing potential or not sexually active)

Exclusion Criteria :

* For a woman of child-bearing potential sexually active, known or suspected pregnancy or positive serum/urine pregnancy test (not applicable for participants aged 2 to 17 years' females not of child-bearing potential or not sexually active)
* Breast-feeding woman
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances
* Chronic illness, at a stage that could interfere with trial conduct or completion, in the opinion of the investigator
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of immune response
* Receipt or planned receipt of any vaccine (other than influenza vaccine which can be given 2 weeks or more before vaccination) in the 4 weeks preceding or following the trial vaccination
* Known Human Immunodeficiency Virus (HIV), Hepatitis B surface (HBs) antigen , or Hepatitis C seropositivity as reported by the participant/parent/guardian and/or based on medical history
* History of documented invasive meningococcal disease
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular vaccination
* Subjects deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent
* Personal or family history of Guillain-Barré Syndrome

Temporary contraindications delaying vaccination until resolved:

* Febrile illness (temperature ≥38.0°C) or moderate or severe acute illness/infection on the day of vaccination
* Received oral or injected antibiotic therapy within the 72 hours prior to any blood draw

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA.
Locations (3):
- India (3):
  - Bangalore
  - Mumbai
  - New Delhi

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 11 June to 01 October 2010 in 3 clinical centers in India.
Pre-assignment Details: A total of 300 participants that met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Age 2 to 11 Years Group: Participants at age 2 to 11 years on enrollment.
- Age 12 to 17 Years Group: Participants aged 12 to 17 years at enrollment.
- Age 18 to 55 Years Group: Participants aged 18 to 55 years at enrollment
Period: Overall Study
Arm/Group | Age 2 to 11 Years Group | Age 12 to 17 Years Group | Age 18 to 55 Years Group
Started | 100 | 100 | 100
Completed | 99 | 98 | 100
Not Completed | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age 2 to 11 Years Group | Age 12 to 17 Years Group | Age 18 to 55 Years Group | Total
Number analyzed (Participants) | 100 | 100 | 100 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100 | 100 | 0 | 200
  Between 18 and 65 years | 0 | 0 | 100 | 100
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 7.2 (3.1) | 14.2 (1.4) | 34.8 (9.2) | 18.7 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 48 | 38 | 139
  Male | 47 | 52 | 62 | 161
Region of Enrollment [Number; unit: Participants]
  India | 100 | 100 | 100 | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Vaccine Antibody Titers at ≥ 8 Before and After Menactra Vaccination
Description: Antibodies to Menactra vaccine were measured by the Serum bactericidal assay baby rabbit complement (SBA BR) Test.
Time Frame: Baseline and 21 days post-vaccination
Population: Menactra vaccine antibody titers were determined in the immunogenicity analysis set.
Measure: Number; unit: Participants
Arm/Group | Age 2 to 11 Years Group | Age 12 to 17 Years Group | Age 18 to 55 Years Group
Number analyzed (Participants) | 100 | 100 | 100
Participants
  Serogroup A (Pre-vaccination; N= 100, 100, 100) | 17 | 27 [0 to 0] | 23 [0 to 0]
  Serogroup A (Post-vaccination; N= 99, 97, 98) | 95 | 94 [0 to 0] | 97 [0 to 0]
  Serogroup C (Pre-vaccination; N= 100, 100, 100) | 24 | 43 [0 to 0] | 66 [0 to 0]
  Serogroup C (Post-vaccination; N= 99, 98, 100) | 91 | 95 [0 to 0] | 99 [0 to 0]
  Serogroup Y (Pre-vaccination; N= 100, 100, 100) | 92 | 92 [0 to 0] | 89 [0 to 0]
  Serogroup Y (Post-vaccination; N= 99, 97, 98) | 99 | 97 [0 to 0] | 98 [0 to 0]
  Serogroup W-135 (Pre-vaccination; N=100, 100, 100) | 54 | 68 [0 to 0] | 52 [0 to 0]
  Serogroup W-135 (Post-vaccination; N= 99, 97, 99) | 96 | 97 [0 to 0] | 99 [0 to 0]

2. Primary Outcome: Serum Bactericidal Assay Baby Rabbit Complement (SBA BR) Geometric Mean Titers Before and Post Menactra Vaccination
Description: Antibodies to Menactra antigens determined by the serum bactericidal assay baby rabbit complement (SBA-BR) test.
Time Frame: Day 0 and Day 30 post-vaccination
Population: Geometric mean titers were determined in the immunogenicity analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution (1/dil)
Arm/Group | Age 2 to 11 Years Group | Age 12 to 17 Years Group | Age 18 to 55 Years Group
Number analyzed (Participants) | 100 | 100 | 100
1/dilution (1/dil)
  Serogroup A (Pre-vaccination; N= 100, 100, 100) | 9.51 [6.43 to 14.1] | 15.0 [9.65 to 23.4] | 9.78 [6.90 to 13.9]
  Serogroup A (Post-vaccination; N= 99, 97, 98) | 1145 [854 to 1536] | 1324 [1002 to 1750] | 2261 [1749 to 2924]
  Serogroup C (Pre-vaccination; N= 100, 100, 100) | 9.92 [7.01 to 14.0] | 17.9 [12.2 to 26.2] | 56.9 [36.6 to 88.3]
  Serogroup C (Post-vaccination; N= 99, 98, 100) | 610 [392 to 949] | 2343 [1563 to 3512] | 7486 [5380 to 10417]
  Serogroup Y (Pre-vaccination; N= 100, 100, 100) | 355 [256 to 491] | 309 [222 to 430] | 156 [110 to 222]
  Serogroup Y (Post-vaccination; N= 99, 97, 98) | 1964 [1607 to 2399] | 3190 [2502 to 4067] | 3926 [2855 to 5398]
  Serogroup W-135 (Pre-vaccination; N=100, 100, 100) | 31.3 [20.6 to 47.7] | 47.8 [32.3 to 70.9] | 28.6 [18.6 to 44.1]
  Serogroup W-135 (Post-vaccination; N= 99, 97, 99) | 1756 [1240 to 2486] | 2538 [1947 to 3307] | 3183 [2360 to 4293]

3. Primary Outcome: Percentage of Participants With at Least a 4-fold Increase in Antibodies to Menactra Vaccine Antigens Post Vaccination
Description: Antibodies to Menactra antigens determined by the serum bactericidal assay baby rabbit complement (SBA-BR) test.
Time Frame: Day 0 to 30 post-vaccination
Population: Four-fold antibody increase were determined in the immunogenicity analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Age 2 to 11 Years Group | Age 12 to 17 Years Group | Age 18 to 55 Years Group
Number analyzed (Participants) | 100 | 100 | 100
Percentage of Participants
  Serogroup A (N = 99, 97, 98) | 85 | 85 [0 to 0] | 96 [0 to 0]
  Serogroup C (N = 99, 98, 100) | 88 | 91 [0 to 0] | 96 [0 to 0]
  Serogroup Y (N = 99, 97, 98) | 68 | 75 [0 to 0] | 89 [0 to 0]
  Serogroup W-135 (N = 99, 97, 99) | 93 | 96 [0 to 0] | 97 [0 to 0]

4. Primary Outcome: Number of Participants Reporting a Solicited Injection Site or Systemic Reactions Following Menactra Vaccination
Description: Solicited injection site: Pain, Erythema (Redness), and Swelling. Solicited Systemic reaction: Fever (Temperature), Headache, Malaise, and Myalgia
Time Frame: Day 0 to 7 post-vaccination
Population: Safety parameters were assessed in the safety analysis set
Measure: Number; unit: Participants
Arm/Group | Age 2 to 11 Years Group | Age 12 to 17 Years Group | Age 18 to 55 Years Group
Number analyzed (Participants) | 100 | 100 | 100
Participants
  Any Solicited injection site pain | 30 | 23 [0 to 0] | 38 [0 to 0]
  Grade 3 pain (Incapacitating) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Any Solicited injection site erythema | 7 | 1 [0 to 0] | 0 [0 to 0]
  Grade 3 erythema (≥5 cm [2-11 years] or >10 cm) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Any Solicited injection site swelling | 10 | 4 [0 to 0] | 0 [0 to 0]
  Grade 3 swelling (≥5 cm [2-11 years] or >10 cm) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Any Solicited fever | 11 | 3 [0 to 0] | 5 [0 to 0]
  Grade 3 fever (≥ 39.0°C) | 3 | 2 [0 to 0] | 2 [0 to 0]
  Any Solicited headache | 12 | 19 [0 to 0] | 19 [0 to 0]
  Grade 3 headache (significant) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Any Solicited malaise | 9 | 13 [0 to 0] | 5 [0 to 0]
  Grade 3 malaise (significant) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Any Solicited myalgia | 13 | 8 [0 to 0] | 12 [0 to 0]
  Grade 3 myalgia (significant) | 0 | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination (Day 0) to up to 6 months post vaccination
Arm/Group | Age 2 to 11 Years Group | Age 12 to 17 Years Group | Age 18 to 55 Years Group
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 30/100 | 23/100 | 38/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age 2 to 11 Years Group (N=100) | Age 12 to 17 Years Group (N=100) | Age 18 to 55 Years Group (N=100)
Fever (General disorders) | 11 (11) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 12 (12) | 19 (19) | 19 (19)
Malaise (General disorders) | 9 (9) | 13 (13) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 8 (8) | 12 (12)
Injection site pain (General disorders) | 30 (30) | 23 (23) | 38 (38)
Injection site erythema (General disorders) | 7 (7) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 10 (10) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.